CLINICAL TRIAL: NCT05286385
Title: A Pre-Marketing, Prospective, Single-Site, Open-Label, Within-Subject, Pilot, Interventional Study of Adult Cochlear Implant Speech Perception With the CP1150 Sound Processor Compared With the Next Generation of Signal Processing Technology
Brief Title: CP1150 Sound Processor Speech Perception Compared With the Next Generation of Signal Processing Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CLTD5818
Record Dates: First submitted 2022-02-22; First posted 2022-03-18 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-02

CONDITIONS: Hearing Impairment, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test Order 1 (Experimental): CP1150, then CP1150 NF, then CP1110, then CP1150 + FF
  Interventions: Device: CP1150 Sound Processor; Device: CP1150 NF; Device: CP1150 + FF; Device: CP1110
- Test Order 2 (Experimental): CP1150 NF, then CP1150 + FF, then CP1150, then CP1110
  Interventions: Device: CP1150 Sound Processor; Device: CP1150 NF; Device: CP1150 + FF; Device: CP1110
- Test Order 3 (Experimental): CP1150 + FF, then CP1110, then CP1150 NF, then CP1150
  Interventions: Device: CP1150 Sound Processor; Device: CP1150 NF; Device: CP1150 + FF; Device: CP1110
- Test Order 4 (Experimental): CP1110, thenCP1150, then CP1150 + FF, then CP1150 NF
  Interventions: Device: CP1150 Sound Processor; Device: CP1150 NF; Device: CP1150 + FF; Device: CP1110

INTERVENTIONS:
Device: CP1150 Sound Processor — Speech perception tests whilst the subject is fitted with the CP1150 Sound Processor
Device: CP1150 NF — Speech perception tests whilst the subject is fitted with the CP1150 modified firmware (the addition of notch filters at 978Hz, 1956Hz, 2934Hz, 3912Hz).
Device: CP1150 + FF — Speech perception tests whilst the subject is fitted with the CP1150 Sound Processor with ForwardFocus.
Device: CP1110 — Speech perception tests whilst the subject is fitted with the CP1110 Sound Processor.

SUMMARY:
This clinical study aims to investigate speech performance in quiet with an OTE Sound Processor with modified firmware compared with the commercially available CP1150. The study also investigates CP1110 and CP1150 with Forward Focus.

DETAILED DESCRIPTION:
This study will build on the evidence previously collected on OTE and BTE Sound Processors and will support the design goals for access to the same sound processing algorithms across future OTE and BTE variants, including evidence required on the automation of FF and future implant compatibility.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Post lingually deafened
3. Implanted with the CI600 Series, CI500 Series or Freedom Series
4. At least 6 months experience with a cochlear implant.
5. At least 3 months experience with a CP910/920, CP950, CP1150, or CP1000 Sound Processor
6. MAP Total Stimulation Rate of 7.2kHz or greater
7. Able to score 30% or more with CI alone on a monosyllabic words in quiet test
8. Willingness to participate in and to comply with all requirements of the protocol
9. Fluent speaker in English as determined by the investigator
10. Willing and able to provide written informed consent

Exclusion Criteria:

1. Additional disabilities that would prevent participation in evaluations.
2. Implant location that would result in undesirable hearing performance or discomfort with an off-the-ear sound processor, as determined by the investigator.
3. Unable or unwilling to comply with the requirements of the clinical investigation, as determined by the Investigator.
4. Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
5. Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation.
6. Currently participating or participated in another interventional clinical study/trial in the past 30 days unless (if less than 30 days) the prior investigation was Cochlear sponsored and determined by the investigator to not impact clinical findings of this investigation.
7. Implanted with other active implantable medical devices (e.g. pacemaker, defibrillator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cochlear Sydney, Macquarie Park, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants (CP1150 SP Compared With Next Generation Signal Processing Technology): All study participants attended a single study visit. At the study visit, subjects underwent hearing assessments. Speech perception tests were carried out in all participants in a randomized manner with 4 interventions involving the CP1150 Sound Processor, CP1150 with modified firmware, CP1150 Sound Processor with Forward Focus and the CP1110 Sound Processor
Period: Overall Study
Arm/Group | All Study Participants (CP1150 SP Compared With Next Generation Signal Processing Technology)
Started | 10
CP1150 Sound Processor | 10
CP1150 Sound Processor With Modified Firmware | 10
CP1150 Sound Processor With Forward Focus | 10
CP1110 Sound Processor | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants (CP1150 SP Compared With Next Generation Signal Processing Technology): All study participants attended a single study visit. At the study visit, subjects underwent hearing assessments. Speech perception tests were carried out in all study participants in a randomized manner with 4 interventions involving the CP1150 Sound Processor, CP1150 with modified firmware, CP1150 Sound Processor with Forward Focus and the CP1110 Sound Processor.
Arm/Group | All Study Participants (CP1150 SP Compared With Next Generation Signal Processing Technology)
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 70.6 [58 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 10
Age at hearing implant [Mean (Standard Deviation); unit: years] | 59.2 (7.64)

OUTCOME MEASURES:

1. Primary Outcome: Speech Perception in Quiet Using an CP1150 Sound Processor
Description: Paired difference in percentage CNC Words correct in quiet with the CP1150 Sound Processor and CP1150 Sound Processor with modified firmware.
Time Frame: One day (in booth testing)
Measure: Mean (Standard Deviation); unit: percentage of correct words
Groups:
- CP1150 NF: All subjects tested with CP1150 Sound Processor with modified firmware.
- CP1150: All subjects test with CP1150
Arm/Group | CP1150 NF | CP1150
Number analyzed (Participants) | 10 | 10
percentage of correct words | 13.82 (10) | 11.53 (10)
Statistical Analysis 1: Comparison: CP1150 NF vs CP1150; Test type: Non-Inferiority — Non-inferiority margin -10%; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-6.29 to 0.29], Standard Deviation 4.59

2. Secondary Outcome: Speech Perception in Quiet Using CP1150 Sound Processor Using Forward Focus Combined With Standard Microphone Directionality.
Description: Paired difference in percentage CNC Words correct in quiet with the CP1150 Sound Processor and CP1150 Sound Processor with forward focus
Time Frame: One day (in booth testing)
Measure: Mean (Standard Deviation); unit: percentage of correct words
Groups:
- CP1150 + FF: All subjects tested with CP1150 Sound Processor with forward focus
- CP1150: All subjects tested with the CP1150 Sound Processor
Arm/Group | CP1150 + FF | CP1150
Number analyzed (Participants) | 10 | 10
percentage of correct words | 11.24 (10) | 11.53 (10)
Statistical Analysis 1: Comparison: CP1150 + FF vs CP1150; Test type: Non-Inferiority — Non-inferiority margin -10%; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-8.04 to 3.44], Standard Deviation 8.03

3. Secondary Outcome: Speech Perception in Quiet With CP1150 and CP1110 Sound Processors
Description: Paired difference in percentage CNC Words correct in quiet with the CP1150 Sound Processor and CP1110 Sound Processor
Time Frame: One day (in booth testing)
Measure: Mean (Standard Deviation); unit: percentage of correct words
Groups:
- CP1150: All subjects tested with CP1150 Sound Processor
- CP1110: All subjects tested with the CP1110 Sound Processor
Arm/Group | CP1150 | CP1110
Number analyzed (Participants) | 10 | 10
percentage of correct words | 11.53 (10) | 11.97 (10)
Statistical Analysis 1: Comparison: CP1150 vs CP1110; Test type: Non-Inferiority — Non-inferiority margin -10%; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-2.95 to 3.55], Standard Deviation 4.55

ADVERSE EVENTS:
Time Frame: 1 day (in booth testing)
Description: Speech perception tests were carried out in all study participants in a randomized manner with 4 interventions involving the CP1150 Sound Processor, CP1150 sound processor with modified firmware, CP1150 Sound Processor with Forward Focus and the CP1110 Sound Processor. All study participants attended a single study visit. At the study visit safety was assessed by recording and summarizing all adverse events and no adverse events were observed during the speech perception tests.
Groups:
- Test Orders 1, 2, 3 & 4 Combined: All subjects tested regardless of order of testing.
Arm/Group | Test Orders 1, 2, 3 & 4 Combined
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT05286385/Prot_002.pdf
  • Statistical Analysis Plan (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT05286385/SAP_001.pdf